CLINICAL TRIAL: NCT06255132
Title: Exploratory Study on the Role of Automated Pupillometry in Patients Underwent Cardiac Surgery to Predict Postoperative Delirium
Brief Title: Automated Pupillometry in Patients Underwent Cardiac Surgery to Predict Postoperative Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4079CESC
Record Dates: First submitted 2023-10-26; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Delirium
Keywords: automated pupillometry; cardiac surgical procedures
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients undergoing open heart surgery (Experimental)
  Interventions: Device: Automated pupillometer NPi-200

INTERVENTIONS:
Device: Automated pupillometer NPi-200 — Pupillary variables in both eyes are recorded and measured with NPi-200 every 30 minutes from the induction of anesthesia. At the end of the surgery, the patient is transferred to the intensive care unit (ICU), and the pupillary variables are recorded until the patient regains consciousness (Richmond agitation sedation scale, RASS>-3). Specific hemodynamic, respiratory, surgical, and EBP data are also recorded as well as NIRS variables.
  As soon as the patient had regained consciousness (RASS > 3), they were assessed for delirium for a total period of five days. Nursing and/or medical staff administered the CAM-ICU score to patients twice a day (morning and afternoon).

SUMMARY:
The rate of postoperative delirium in patients who underwent cardiac surgery is very high. Different predictors and/or scores were studied for the prediction of Post Operative Delirium (POD)after heart surgery, but none of them was validated. The investigators aim to explore the role of pupillary alterations during anesthesia in open-heart surgery.

The goal of this prospective study is to evaluate if pupil alterations during cardiac surgery, evaluated by an automated pupillometer (NPi-200) ( AP), could predict postoperative delirium.

DETAILED DESCRIPTION:
Consent was obtained during the hospitalization before the planned surgery.

On the day of surgery, before general anesthesia is started, Near-infrared spectroscopy (NIRS) sensors are applied to the patient's forehead bilaterally and the baseline value is recorded. Pupils' variables (i.e., diameter, % constriction, constriction velocity, dilation velocity, latency, NPi) are also recorded from both the right and left eye with AP (NPi-200).

From the induction of anesthesia, pupillary variables in both eyes are recorded and measured every 30' such as the concomitant NIRS values (at least one measurement per eye per operative phase). Moreover, hemodynamic and respiratory parameters concomitant with the pupillary measurements are measured.

Following surgery, the patient is transferred to the Cardiac Intensive Care Unit. There, NIRS monitoring as as well as automated pupillometry measurements will be maintained until the patient regains consciousness (defined as RASS sedation scale >-3).

Once the patient has regained consciousness (RASS>-3), is assessed twice a day (morning and afternoon) with the Confusion assessment method-intensive care unit (CAM-ICU) score by the nursing staff and/or medical staff. The presence or absence of POD will then be reported as well as any pharmacological and non-pharmacological treatments.

Any neurological complications and diagnostic investigations arising in the post-operative period will also be noted.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective open cardiac surgery (>18 yr)
* Elective open cardiac surgery and cardiopulmonary bypass

Exclusion Criteria:

* Patients <18 years of age
* Emergency surgeries
* Heart operations, not including extracorporeal circulation
* Surgery for aortic arch dissection with hypothermia and/or circulatory arrest
* Patients affected by psychiatric disorders undergoing with or without neuroleptic therapy
* Patients who have the refused consent
* Patients with ocular problems (acute or previous trauma to one or both eyes, blindness, ocular prosthesis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Correlation between neurological pupil index (NPi) and Post-operative delirium | Intraoperative (day 0)
  We want to relate pupillary reactivity, assessed with automated pupillometry such as the Neurological pupil index (numerical value:0-5) during surgery, with Postoperative delirium (assessed with CAM-ICU score during the first 5 postoperative days).

SECONDARY OUTCOMES:
Correlation between early prediction model for delirium (E-PRE-DELIRIC) and POD | E-PREDELIRIC is calculated at ICU admission ( day 0)
  E-PREDELIRIC is a standard prediction model for ICU delirium (%) and is calculated at ICU admission. We aim to evaluate the correlation between the model and Postoperative delirium in cardiovascular patients
Correlation between regional cerebral saturation (rSO2) and POD occurrence | rSO2 is monitored during surgery (Day 0)
  Regional cerebral saturation (rSO2) ranges between 0 and 100% and is a standard of care during open heart surgery. We want to evaluate the correlation between intraoperative cerebral saturation during surgery and POD.
Correlation between Cardiopulmonary bypass duration and POD. | Intraoperative
  Cardiopulmonary bypass duration within heart surgery is variable (min), depending on different surgical factors. We aim to evaluate if the duration of CPB could be related to POD occurrence
Multivariate model for POD prediction. | Day 0
  a multivariate analysis will be performed to build a prediction model for postoperative delirium in the specific population of cardiovascular patients who underwent open heart surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Gottin, Prof., Study Director — Universita di Verona; Federico Romagnosi, MD, Principal Investigator — Universita di Verona
Locations (1):
- Unit of Cardiothoracic Anesthesia and Intensive Care, University hospital of Verona, Verona, Vr, Italy